CLINICAL TRIAL: NCT04050124
Title: Impact of Promogran Prisma™ on Pain of Split-thickness Skin Graft Donor Sites Compared to Standard of Care Alone
Brief Title: Impact of Prisma on Donor Site Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19-00437
Record Dates: First submitted 2019-08-07; First posted 2019-08-08 (Actual); Results first posted 2024-04-16 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-03

CONDITIONS: Skin Graft Disorder; Donor Site Complication
Keywords: Donor site pain after skin graft harvesting
MeSH Terms: interventions — Bandages

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Promogran Prisma (Experimental): Following standard of care split thickness skin grafting, patients randomized to the intervention group will receive Promogan Prisma as the primary contact dressing at the donor grafting site.
  Interventions: Device: Promogran Prisma; Device: Standard of care (SOC) dressings
- Standard of care (SOC) dressings (Active Comparator)
  Interventions: Device: Standard of care (SOC) dressings

INTERVENTIONS:
Device: Promogran Prisma — Promogran+SOC; composite collagen, silver-oxidized regenerated cellulose matrix
  Arms: Promogran Prisma
Device: Standard of care (SOC) dressings — standard of care dressing on donor site pain for patients undergoing split-thickness skin grafting in preparation for a larger study.

SUMMARY:
The purpose of this study is to assess the feasibility of evaluating the use of a composite collagen, silver-oxidized regenerated cellulose matrix compared to the standard of care dressing on donor site pain for patients undergoing split-thickness skin grafting in preparation for a larger study.

ELIGIBILITY:
Inclusion Criteria:

* Patient scheduled to undergo STSG for any reason
* Patient, or designated healthcare proxy, has read and signed the IRB-approved informed consent form.

Exclusion Criteria:

* Active infection or history of radiation to the donor site
* Patient has a known sensitivity to Promogran Prisma™ or silver
* Elevated INR >3.0
* Insensate at the donor site
* Chronic narcotic use (>6 months of daily use)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2019-11-07 (Actual); Primary Completion 2021-11-29 (Actual); Study Completion 2021-11-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Gorenstein, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Promogran Prisma | Standard of Care (SOC) Dressings
Started | 8 | 9
Completed | 7 | 9
Not Completed | 1 | 0
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Promogran Prisma | Standard of Care (SOC) Dressings | Total
Number analyzed (Participants) | 7 | 9 | 16
Age, Continuous [Mean (Full Range); unit: years] | 70.5 [38 to 92] | 69.55 [53 to 84] | 69.88 [38 to 92]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 5 | 7
  Male | 5 | 4 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 7 | 9 | 16
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 6 | 6
  White | 6 | 3 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 9 | 16

OUTCOME MEASURES:

1. Primary Outcome: Pain Score on Visual Analogue Scale (VAS)
Description: Pain score is measured using a VAS ranging from 0-10, where 0 = no pain and 10 = unbearable pain. Participants select the number that best reflects their current status. The total score is the numerical response; lower scores indicate lower pain.
Time Frame: Postoperative Day 1
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Promogran Prisma | Standard of Care (SOC) Dressings
Number analyzed (Participants) | 7 | 9
score on a scale | 2 [0 to 8] | 2 [0 to 8]

ADVERSE EVENTS:
Time Frame: 6 weeks
Description: non- systematic: self report and clinical assesment on weekly clinic visits
Arm/Group | Promogran Prisma | Standard of Care (SOC) Dressings
All-Cause Mortality (participants affected / at risk) | 1/8 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/9
Other Adverse Events (participants affected / at risk) | 0/8 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-15): https://cdn.clinicaltrials.gov/large-docs/24/NCT04050124/Prot_SAP_000.pdf